CLINICAL TRIAL: NCT01345591
Title: Structural Fat Grafting for Craniofacial Trauma
Brief Title: A Study to Evaluate the Results of Facial Soft Tissue Reconstruction in Patients Who Have Suffered Traumatic Injury
Acronym: BTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO09060101
Record Dates: First submitted 2011-04-14; First posted 2011-05-02 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Facial Injuries; Adipose Tissue
Keywords: BTI; Craniomaxillofacial (CMF) Battle-injured (BI); Facial Trauma; Fat Grafts; Autogenous Fat Transfers (AFT); Wounded warriors
MeSH Terms: conditions — Facial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fat Grafting (Experimental): Twenty (20) subjects who have had severe facial trauma, 18 years of age and older enrolled to clinical trial will receive Fat grafting intervention procedure
  Interventions: Procedure: Fat Grafting

INTERVENTIONS:
Procedure: Fat Grafting

SUMMARY:
Injuries resulting in facial trauma are common, and can have devastating consequences on your quality of life. While the facial bones can often be reconstructed, physicians strive to find better ways to accurately restore injured facial features.

In this clinical trial funded by the Department of Defense, the investigators are evaluating how effectively fat grafting can restore facial features, and how the filling effect of the fat graft lasts over time in participants with visible facial injuries. All procedures for this research study will be performed at the University of Pittsburgh Medical Center.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate how well the filling effect of the fat remains over time. A person's own fat may be used to improve the appearance of the body by moving it from an area where it is less needed. This is called fat grafting, and it is a common procedure, performed approximately 65,000 times by plastic surgeons in the United State last year. The fat is usually taken from the thighs or abdomen with a small liposuction tube and then moved to an area that has lost volume or fullness due to aging, trauma, surgery, birth defects, or other causes. Typically, the transferred fat results in an increase in volume of the body site being treated.

Fat grafting is a minimally invasive surgical procedure in which a person's own fat may be used to improve the appearance of the body by moving it from an area where it is less needed. The fat is usually taken from the thighs or abdomen with a small liposuction tube and then moved to an area that has lost shape or fullness due to injury. This procedure is performed through very small incisions that allow a hollow tube to pass through.

Fat grafting is a common cosmetic and reconstructive procedure. It was performed approximately 65,000 times by plastic surgeons in the United States last year. Typically, the transferred fat results in an increase in volume and shape of the body site being treated. The investigators believe this clinical technique of fat grafting could be of significant benefit to patients with facial injuries. The fat grafting procedure being performed in this trial is considered to be research, but not an experimental procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and able to provide informed consent
2. Have suffered injury resulting in craniofacial volume defects which could be treated with a graft volume of between 5 and 150 cc of lipoaspirate
3. Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved
4. Volume defects are covered by intact skin and do not communicate with oral cavity or sinuses
5. The three dimensional geometry of the volume defects would allow for treatment with lipoaspirate injection that in a manner that at least two distinct treated areas could be discerned on gross examination and radiographically (e.g. treated regions are on opposite sides of the face, on lower face versus upper face, or separated by a bony landmark such as zygoma. This would include the ability to treat an uninjured contralateral region with lipoaspirate in order to obtain symmetry.
6. Willing and able to comply with follow up examinations, including radiographic studies -

Exclusion Criteria:

1. Age less than 18 years
2. Inability to provide informed consent
3. Craniofacial defects intended for treatment have open wounds or communicate with oral cavity or sinus (note: presence of such a defect in the setting of another defect(s) that meets treatment criteria will not exclude the patient from participating).
4. Active infection anywhere in the body
5. Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
6. Known coagulopathy
7. Pregnancy -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Rubin, MD, Principal Investigator — Associate Professor of Plastic Surgery at the University of Pittsburgh, Faculty appointment-McGowan Institute of Regenerative Medicine
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is the Principal Investigator's intention to make stored samples and subject information de-identified available to secondary investigators (investigators not listed on the front page of this consent document) after all research study testing has been completed. These stored samples and associated subject information will not include subject identifiers.

REFERENCES:
- [Background] Coleman SR. Structural fat grafting: more than a permanent filler. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):108S-120S. doi: 10.1097/01.prs.0000234610.81672.e7. PMID 16936550
- [Background] Burnouf M, Buffet M, Schwarzinger M, Roman P, Bui P, Prevot M, Deleuze J, Morini JP, Franck N, Gorin I, Dupin N. Evaluation of Coleman lipostructure for treatment of facial lipoatrophy in patients with human immunodeficiency virus and parameters associated with the efficiency of this technique. Arch Dermatol. 2005 Oct;141(10):1220-4. doi: 10.1001/archderm.141.10.1220. PMID 16230558
- [Background] Kaufman MR, Bradley JP, Dickinson B, Heller JB, Wasson K, O'Hara C, Huang C, Gabbay J, Ghadjar K, Miller TA. Autologous fat transfer national consensus survey: trends in techniques for harvest, preparation, and application, and perception of short- and long-term results. Plast Reconstr Surg. 2007 Jan;119(1):323-331. doi: 10.1097/01.prs.0000244903.51440.8c. PMID 17255689

RESULTS

PARTICIPANT FLOW:
Groups:
- Fat Grafting: fat grafting for facial trauma
Period: Overall Study
Arm/Group | Fat Grafting
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fat Grafting
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
volume [Mean (Standard Deviation); unit: milliliters] | 1.0 (0.0001)
tissue thickness [Mean (Standard Deviation); unit: milliliters] | 0.352 (0.180)

OUTCOME MEASURES:

1. Primary Outcome: Volume
Description: fat graft volume
Time Frame: 3 months and 9 months post op.
Measure: Mean (Standard Deviation); unit: milliliters
Groups:
- Fat Graft Volume at 3 Months: fat grafting for facial trauma, volume measured at 3 months post-op
- Fat Graft Volume at 9 Months: fat grafting for facial trauma, volume measured at 9 months post-op
Arm/Group | Fat Graft Volume at 3 Months | Fat Graft Volume at 9 Months
Number analyzed (Participants) | 19 | 19
milliliters | 0.576 (0.188) | 0.621 (0.191)

2. Secondary Outcome: SWAP, COPE and CSQ-8
Description: three questionnaires were evaluated: 1) SWAP (satisfaction with appearance scale) is a psychological test for personality diagnosis and clinical case formulation; 14 questions are asked on a scale of 0-7 where 7 indicates descriptive of the subjects and 0 is irrelevant to the subject for a total score range of 0-98. 2) COPE scale assesses a broad range of coping responses over 28 questions scaled from 1-4 with a total score range of 28-112 where the higher score indicates higher frequency of coping mechanisms used by the subject. 3) CSQ-8 assesses patient satisfaction with the treatment through 8 questions ranked 1-4 on a total scale from 8-32 where higher scores indicate greater satisfaction.
Time Frame: as assessed at baseline, 7-21 days, 3 months and 9 months post op.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fat Grafting_evaluation at Baseline: quality of life measurement at baseline to include SWAP, COPE and CSQ-8 questionnaires
- Fat Grafting_7-21 Days Post op: quality of life measurement at 7-21 days post-op to include SWAP, COPE and CSQ-8 questionnaires
- Fat Grafting_3 Months Post op: quality of life measurement at 3 months post-op to include SWAP, COPE and CSQ-8 questionnaires
- Fat Grafting_9 Months Post-op: quality of life measurement at 9 months post-op to include SWAP, COPE and CSQ-8 questionnaires
Arm/Group | Fat Grafting_evaluation at Baseline | Fat Grafting_7-21 Days Post op | Fat Grafting_3 Months Post op | Fat Grafting_9 Months Post-op
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale
  SWAP | 59.7 (11.1) | 57.8 (7.0) | 57.9 (8.3) | 56.3 (6.3)
  COPE | 57.1 (8.5) | 56.8 (13.1) | 54.4 (13.5) | 55.1 (7.7)
  CSQ-8 | 27.0 (2.9) | 30.9 (2.4) | 31.3 (2.2) | 30.7 (2.4)

ADVERSE EVENTS:
Arm/Group | Fat Grafting
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fat Grafting (N=20)
bruising (Surgical and medical procedures) | 20
swelling at injection site (Surgical and medical procedures) | 20
warmth (Vascular disorders) | 20
redness at injection site (Surgical and medical procedures) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes